CLINICAL TRIAL: NCT00393770
Title: A Pilot Study to Evaluate the Short-term Effects of Acetyl-carnitine on Insulin Resistance and the Metabolic Syndrome in Patients at Increased Risk of Type 2 Diabetes: Acetyl-carnitine in Insulin Resistance
Brief Title: Acetylcarnitine and Insulin Sensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Norberto Perico, Mario Negri Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAC01
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Risk of type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acetylcarnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-acetylcarnitine (Experimental)
  Interventions: Drug: L-acetylcarnitine

INTERVENTIONS:
Drug: L-acetylcarnitine — 250-500 mg/kg/die.

SUMMARY:
Decreased insulin sensitivity (e.g. insulin resistance) is a hallmark and a major pathogenic factor of type 2 diabetes. It is the key factor of the metabolic syndrome - a cluster of arterial hypertension, obesity, impaired glucose tolerance, dyslipidemia, coagulation abnormalities,albuminuria and increased cardiovascular risk - that may precede or accompany type 2 diabetes.

Insulin function and the abnormalities associated with insulin resistance, may have a major role in preventing type 2 diabetes and, in the long-term, diabetes micro- and macrovascular complications. Carnitine is involved in lipids and carbohydrates metabolism and acetyl-L-carnitine(ALC), an intramitochondrial carrier of acylic group, may modulate cell fuel substrate utilization. Studies found that carnitine may improve insulin sensitivity and glucose disposal in healthy subjects and in patients with type 2 diabetes. A recent study also found that a primed constant infusion of acetyl-L-carnitine (ALC) may increase glucose utilization in type 2 diabetic patients, possibly restoring the glycogen synthase activity.

Thus, we designed the Acetylcarnitine in insulin resistance study, a pilot, sequential,longitudinal study aimed to assess whether acetyl-carnitine may improve insulin function and lipid profile in patients at increased risk of type 2 diabetes.

DETAILED DESCRIPTION:
Decreased insulin sensitivity (e.g. insulin resistance) is a hallmark and a major pathogenic factor of type 2 diabetes. Diabetes often is related to a cluster of arterial hypertension, obesity, impaired glucose tolerance, dyslipidemia, coagulation abnormalities, albuminuria and increased cardiovascular risk which is called metabolic syndrome. A reduction of insulin-resistance may improve metabolic syndrome, decreasing in the long term the onset of clinical diabetes and the incidence of important cardiovascular and renal complications. In the presence of insulin resistance it is altered the normal signal to the adipose tissue with a consequent reduction of absorption and use of glucose. In subjects with increased fat mass, mainly visceral, it has been shown the influence of several factors, as tumoral necrosis factor alfa (TNF alfa) and fatty free acids (FFAs), on the peripheral activity of the insulin. TNF alfa, a key modulator in fat metabolism, has a direct role on insulin-mediated homeostasis of glucose and fatty acids, regulating the action of lipoprotein lipases and fatty acid carriers influencing CoA synthesis and leptin production that, finally, inhibits insulin secretion by pancreatic beta cells. Increasing of circulating concentration of fatty acids, due to the absence of suppression of lipolysis due to insulin inactivity, contributes to peripheral and hepatic insulin resistance. It is also correlated with a condition of active inflammation, which is linked to a higher incidence of atherosclerosis and cardiovascular risk, typical of diabetes.

Other factors, such as adiponectin and resistin, showed to have a role in glucose metabolism. Adiponectin, a protein produced by adipocytes, has well-known anti-inflammatory and anti-atherogenic actions, and it is postulated to improve insulin sensitivity through the improvement of carbohydrates and lipids metabolism. In contrast, resistin seems to induce insulin resistance and decreased glucose tolerance. Thus, the improvement of metabolic syndrome, by means of an increase of insulin sensitivity and correction of correlated lipids and carbohydrates metabolism may play a primary role in the prevention of type 2 diabetes and, in the long term, may decrease micro- and macro-vascular complications. Large prospective trials will help us to understand cellular mechanisms involved in metabolic syndrome and may be useful to identify new therapeutic targets aimed to reduce insulin resistance. Carnitine is involved in lipids and carbohydrates metabolism and acetyl-L-carnitine (ALC) may increase glucose utilization in type 2 diabetic patients, possibly restoring the glycogen synthase activity. ALC is a mitochondrial carrier of acylic groups, which directly and indirectly participates to carbohydrates metabolism, acting on fatty acids and on glucose oxidation on pyruvate dehydrogenase (PDH). PDH is formed by an enzymatic complex (PDC) which catalyzes an irreversible reaction in carbohydrates oxidation, and it is controlled by a phosphorylation-dephosphorylation cycle, in which Pyruvate Dehydrogenase Kinase uses ATP to phosphorylate PDH causing its inactivation, and Pyruvate Dehydrogenase Phosphatase dephosphorylates PDH inactivating it. Kinase is activated by an increased ratio intramitochondrial acetylCoA/CoA, as we can see in conditions of high fatty acid levels. The consequent reduction of PDC activity, dramatically decreases glucose oxidation. Carnitine participates to trans-esterification, forming acetylcarnitine. By means of catching acylic groups, it decreases ratio acetylCoA/CoA, indirectly stimulating PDC activity and favouring pyruvate oxidation and of glucose. Thus acetylcarnitine can be considered a modulator of substrates utilization in cells, with consequences in the metabolism of both lipids and carbohydrates. Several studies demonstrated that carnitine contributes to the improvement of insulin sensitivity and glucose utilization in both healthy subjects and type 2 diabetics. Thus it is interesting to confirm the hypothesis that acetylcarnitine may improve insulin sensitivity in patients with a risk for type 2 diabetes and verify if this improvement is associated with other components of metabolic syndrome.

Primary aim To evaluate insulin sensitivity (e.g. Glucose disposal rate during an euglycemic hyperinsulinemic clamp) in 40 patients with normal morning fasting glucose and increased risk of type 2 diabetes mellitus.

Secondary aims

* To evaluate drug effects on sitting systolic/diastolic blood pressure, lipid profile, morning fasting glucose and postprandial glucose.
* To assess the correlation between insulin sensitivity and serum inflammatory markers (Erythrocyte Sedimentation Rate, C-reactive protein) and insulin, leptin and adiponectin levels
* To assess treatment tolerability

Design of the study This will be a sequential and longitudinal study.

Potentially eligible patients will have a baseline evaluation of the following parameters:

Clinical Systolic/diastolic blood pressure, Heart rate, Body weight (BW), B.M.I., Total body water (TBW)*, Fat-free mass (FFM) **, Fat mass (FM) *** Metabolic Fasting morning blood glucose; oral glucose tolerance test Insulin, leptin, adiponectin level Lipid profile Total, VLDL and HDL cholesterol, total triglycerides, Apolipoprotein A and B Inflammatory markers Erythrocyte Sedimentation Rate, C-reactive protein and plasma TNF alfa Patients satisfying the inclusion/exclusion criteria will have their insulin sensitivity evaluated by an euglycemic hyperinsulinemic clamp and will enter a six month treatment period with Acetylcarnitine 2 g/day. At the end of the treatment period and 2 months after treatment withdrawal, all baseline parameters, including insulin sensitivity, will then be evaluated. No changes in diet and in concomitant treatments (in particular with diuretics, ACE inhibitors, angiotensin II receptor antagonists, dihydro and non-dihydro calcium channel blockers, statins) will be introduced throughout the whole study period.

* Calculated by the Hume and Weyers formula: TBW in males = (0.2968 x weight in kg) + (0.1948 x height in cm) - 14.0129 TBW in females = (0.1838 x weight in kg) + (0.3446 x height in cm) - 35.2701

** FFM = TBW/0.73

*** FM = BW - FFM

ELIGIBILITY:
Inclusion Criteria:

at least three of these

* Relatives with type 2 diabetes
* Age between 40 and 65 years
* Systolic and diastolic pressure ≥ 140 or ≥90 mmHg respectively
* Body mass index ≥25 for men and ≥24 for women
* Triglycerides ≥200 mg/dl
* Serum creatinine ≤1.5 mg/dl, proteinuria ≤ 0.5g/24h
* Capacity to understand the scope and the risks of the study
* written informed consent

Exclusion Criteria:

* Concomitant treatment with steroids, anti-inflammatory and immunosuppressive drug, and any other drug acting on insulin sensitivity and/or insulin secretion, particularly glitazones and other oral hypoglycemic drug
* Treatment with L-acetylcarnitine in the six months before the study
* Previous or concomitant treatment with metformin
* legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-02; Primary Completion 2006-10 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | At 0,3, 6 and 8 months.

SECONDARY OUTCOMES:
Lipid profile. | At 0,3, 6 and 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Perico, MD, Principal Investigator — Mario Negri Institute
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy

REFERENCES:
- [Derived] Ruggenenti P, Cattaneo D, Loriga G, Ledda F, Motterlini N, Gherardi G, Orisio S, Remuzzi G. Ameliorating hypertension and insulin resistance in subjects at increased cardiovascular risk: effects of acetyl-L-carnitine therapy. Hypertension. 2009 Sep;54(3):567-74. doi: 10.1161/HYPERTENSIONAHA.109.132522. Epub 2009 Jul 20. PMID 19620516